CLINICAL TRIAL: NCT04210011
Title: Enhancing the Resilience of Parents by Understanding Their Perceptions, Behaviour, Attitudes, and Experiences Related to Cancer and Its Treatment of Their Child
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: Parental Resilience
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Parents of Children With Cancer
Keywords: Pediatric oncology; Parental resilience

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to describe the psychosocial well-being and quality of life of Hong Kong Chinese parents of children with cancer with the aim at understanding the needs and concerns of parents, including their perceptions, behaviour, attitudes, and experiences related to cancer and its treatment of their child.

DETAILED DESCRIPTION:
Advances in diagnostic techniques and cancer treatments have yielded remarkable increases in the overall survival rates of children with cancer. Inevitably, however, cancer and its treatments may also have long-term effects on the physical and psychological well-being of children with cancer,

Previous studies revealed that parents play a pivotal role in encouraging their child with cancer to engage in healthy behaviours. It was shown that Chinese parental psychological behaviour and control may influence the psychological well-being of their children. Therefore, a thorough understanding the needs and concerns of Chinese parents, including their perceptions, behaviour, attitudes, and experiences related to the illness of their child is essential to facilitate them to empower their child to fight at every step of the long and difficult cancer journey.

On the other hand, the diagnosis of cancer not only undermines children themselves in physical and psychological, but also it brings overwhelming psychological distress for these children's parents. An increasing number of studies have examined patients' resilience in adaptation to cancer. Assessing resilience in parents of children with cancer is crucial for a thorough understanding of their responses to stress and adversity, which is an essential prerequisite for the design of an appropriate psychological intervention to enhance their resilience and foster the development of their coping mechanisms and positive psychological well-being. Nevertheless, the resilience levels and its influencing factors among parents of children with cancer in Hong Kong have never been studied.. Further qualitative and quantitative analyses are necessary to thoroughly explore the relationships between resilience and its influencing factors from a culturally specific perspective, with the goal of developing interventions to promote resilience that are applicable to the Hong Kong Chinese population.

A sequential mixed methods design will be used with a quantitative study (Phase I) will be first conducted and followed by a qualitative study (Phase II). The reason for that the quantitative findings will provide a general understanding of the psychosocial well-being and quality of life of Hong Kong Chinese parents of children with cancer. The qualitative findings and the analysis will help to explain the quantitative findings by exploring the perceptions, behaviour, attitudes, and experiences related to cancer and its treatment of their child.

ELIGIBILITY:
Inclusion Criteria:

* the primary caregiver, either father or mother,
* ability to speak Cantonese and read Chinese-language materials,
* having a child aged 0-16 years and diagnosed with cancer at some time in the previous month and currently undergoing active treatment

Exclusion Criteria:

* Parents with chronic illness and cognitive or learning disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hong Kong Chinese parents of children with cancer admitted to Hong Kong Children's Hospital are eligible. Study inclusion criteria for parents are as follows: (1) the primary caregiver, either father or mother, (2) ability to speak Cantonese and read Chinese-language materials, (3) having a child aged 0-16 years and diagnosed with cancer at some time in the previous month and currently undergoing active treatment. Parents with chronic illness and cognitive or learning disorders will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Connor-Davidson resilience scale | baseline
  Connor-Davidson resilience scale (CD-RISC) will be used to measure the resilience level of parents having children with cancer. It contains a total of 25 items, which can be divided into 3 subcategories: (1) tenacity, (2) strength, and (3) optimism.The total possible scores of the scale range from 0 to 100, with a higher score indicating greater resilience.

SECONDARY OUTCOMES:
The EuroQoL 5-Dimension 5-level | baseline
  The EuroQoL 5-Dimension 5-level (EQ-5D-5L) will be used to measure parents' quality of life.Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
The Center for Epidemiologic Studies Depression Scale (CES-D) | baseline
  The Center for Epidemiologic Studies Depression Scale (CES-D) consists of 20 items, which was originally designed to measure depressive symptoms in general population surveys.Subjects are asked to rate the frequency of each symptom during the past week on a four-point Likert scale representing 'rarely (less than 1 day)', 'some (1-2 days)', 'occasionally (3-4 days)' and 'most (5-7 days)', which are scored from 0 to 3, with total possible scores ranging from 0 to 60. Higher scores indicate a greater risk of depression.
The Chinese version of the State Anxiety Scale for Adults (C-SAS-A) | baseline
  The state anxiety level of parents will be measured by using the The Chinese version of the State Anxiety Scale for Adults (C-SAS-A). The scale consists of 20 items, which are scored from 1 to 4, with possible scores ranging from 20 to 80.
The Multidimensional Scale of Perceived Social Support (MSPSS) | baseline
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item scale with a seven-point scale (from 1=strongly disagree to 7=strongly agree) measuring three sources of support, namely, Family, Friends, and Significant Other.
Parents' perceptions, behaviour, attitudes, and experiences related to the cancer and its treatment of their child | baseline
  Parents will be asked their perceptions, behaviour, attitudes, and experiences related to the cancer and its treatment of their child in the semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong